CLINICAL TRIAL: NCT07313423
Title: Sea Buckthorn Aqueous Infusion Impact on Body Composition Metrics Among Overweight Female Adults.
Brief Title: Sea Buckthorn Aqueous Infusion Impact
Acronym: Sbaii
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Veterinary and Animal Sciences, Lahore - Pakistan (Other)
Responsible Party: Principal Investigator, Qaisar Raza, Assistant professor, University of Veterinary and Animal Sciences, Lahore - Pakistan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UVAS2
Record Dates: First submitted 2025-12-17; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Body Compostition
Keywords: sea buckthorn; aqueous infusion; body composition

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned into two groups in a 1: 1 ratio to either the treatment group (sea buckthorn aqueous infusion) or control group (placebo), both groups will be followed concurrently for 12 weeks to assess changes in bmi, body weight, visceral fat and waist-hip ratio.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Placebo Comparator): The participants in the control group will consume placebo that will match in appearance to the supplement and is used to maintain blinding. Participants will consume freshly prepared sea buckthorn aqueous infusion daily for 12 weeks.
  Interventions: Dietary Supplement: Sea buckthorn aqueous infusion
- 2 (Experimental): Drug (Sea buckthorn aqueous infusion) The participants will consume Sea buckthorn aqueous infusion supplementation daily for 12 weeks. it will be prepared by using 5g sb powder in 250 ml of water.
  Interventions: Dietary Supplement: Sea buckthorn aqueous infusion

INTERVENTIONS:
Dietary Supplement: Sea buckthorn aqueous infusion — Sea buckthorn aqueous infusion prepared by using 5g powder in 250 ml water.

SUMMARY:
* A total of 60 overweight women (BMI 25-29.9 kg/m²), aged 18-50years, will be enrolled and randomized equally into intervention and control groups. The intervention group will consume a 5 g freshly prepared seabuckthorn aqueous infusion daily for 12 weeks, while controls maintain usual habits without supplementation.
* The seabuckthorn aqueous infusion will be prepared by using 250mL of potable boiled water and then cooled to a lukewarm temperature (around 40-45°C). At this point, 5 g of seabuckthorn powder will be added, stirred thoroughly until fully dispersed, and consumed immediately. The infusion will be freshly prepared once daily and administered in the morning after breakfast.

Measurements will be conducted using the InBody 270, a validated bioelectrical impedance analyzer employed in this study to obtain accurate assessments of body weight, body mass index (BMI), waist-hip ratio, and visceral fat levels. The device offers segmental analysis and visceral fat estimation through non-invasive, standardized procedures, ensuring consistency and reliability in longitudinal tracking.

DETAILED DESCRIPTION:
Background: Overweight and obesity have become major public health challengesdisproportionately affecting adult women worldwide, including Pakistan. Functional foodsare gaining attention for their preventive and therapeutic potential, with Sea buckthornemerging as a promising option due to its rich bioactive composition which exhibit antioxidant, anti-inflammatory, and lipid-regulating properties. This research, therefore, seeks to evaluate the effects of sea buckthorn consumption on female body composition, exploring its role as a nutritional intervention for weight management and metabolic health. Hypothesis: Participants consuming sea buckthorn aqueous infusion showsignificant declines in BMI, body weight, visceral fat, and waist-hip ratio. Methodology : A total of 60 overweight women (BMI 25-29.9 kg/m²), aged 18-50years, will be enrolled and will be randomly allocated to intervention and control groups. Theintervention group will consume freshly prepared seabuckthorn aqueous infusion dailyfor12 weeks, while controls maintain usual habits without supplementation. Data analysis : Data will be analyzed using SPSS version 25. Baseline characteristicsbetween groups will be compared using Descriptive statistics (mean ± SD) as appropriate. Between-group comparisons differences will be analyzed using ANOVA. Statistical significance will be set at p < 0.05. Outcome : Supplementation with seabuckthorn aqueous infusion over a 12-weekperiodwill result in notable improvements in body composition measures among overweight female adults.

ELIGIBILITY:
Inclusion criteria females, age 18-50, bmi greater or equal to 25. exclusion criteria current pregnancy or lactation, a history of chronic metabolic or gastrointestinal diseases, use of weight management drugs or supplements, known allergies to sea buckthorn or other documented intolerances, smoking or alcohol consumption, a physical activity level exceeding 1.4, and prior participation in weight loss research programs

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Body weight | 12 weeks
  unit of measurement in kilograms will be measured by weight machine
Body mass index | at the end of intervention (12 week)
  body mass index will be measured using body mass index calculator

SECONDARY OUTCOMES:
visceral fat | at the end of intervention period (12 week)
  visceral fat will be measured using bioelectric impedance analysis
waist-hip ratio | at the end of intervention period ( 12 week)
  waist hip ratio will be measured using measuring tape

CONTACTS AND LOCATIONS:
Locations (1):
- University of veterinary and animal sciences, Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No